CLINICAL TRIAL: NCT04097951
Title: A Randomized, Open-label, Single-dose Study to Evaluate the Safety and the Pharmacokinetics After Oral Concurrent Administration of HDDO-18011 and HDDO-18012 in Healthy Adult Subjects
Brief Title: HDDO-1801 Intervention Trial
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hyundai Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HT-012-01
Record Dates: First submitted 2019-09-17; First posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Respiratory Disease
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Montelukast (Experimental)
  Interventions: Drug: Combinations
- Bepotastine (Experimental)
  Interventions: Drug: Combinations
- Montelukast + Bepotastine (Experimental)
  Interventions: Drug: Combinations

INTERVENTIONS:
Drug: Combinations — Montelukast and Bepotastine Combination

SUMMARY:
A randomized, open-label, single-dose, 3-period, 6-sequence, 3-way crossover study

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male aged 19 years and younger than 50 years old at the time of the screening
2. Those who weigh more than 50 kg and whose calculated BMI is within the 18.0-29.0 kg/m2 range BMI = (weight [kg])/(key [m])2
3. A person who is judged to be suitable for a test through physical examination and examination according to this test plan. That is, a person who has no congenital or chronic diseases and who has not had any pathological symptoms or findings within the last 3 years
4. A person who is judged to be suitable for a test in accordance with this test plan (if the results of a clinical laboratory test are within or outside the reference value of the hospital affiliated with Inha University Medical Center, the tester determines that there is no clinical significance)
5. After hearing the detailed description of this clinical trial and fully understanding it, the person who agrees in writing to decide his/her participation and to comply with the precautions

Exclusion Criteria:

1. Persons with clinical significant cardiovascular, respiratory, liver, kidney, nervous system, endocrine, blood and tumor, mental illness, and urinary tract
2. Persons with gastrointestinal relationship diseases (such as gastrointestinal ulcers, gastritis, gastrointestinal tract diseases, Crohn's disease, etc.) that may affect the absorption of clinical trial medications, and persons with past history of gastrointestinal relationship surgery (except for simple appendectomy or hernia surgery)
3. Those with genetic problems such as galactose intolerance, Lapp lactase deficient or glucose-galactose malabsorption
4. A person with a history of hypersensitivity or clinically significant hypersensitivity to a drug or other drug (aspirin, antibiotics, etc.) that contains the components of Montelukast and the components of Bepotastine or the same family.
5. A person who showed a clinically significant low blood pressure (hydraulic < 90mmHg) or high blood pressure (hydraulic ≥ 150mmHg or dilatant blood pressure ≥ 95mmHg) during the screening test
6. One of the following results is displayed in a screening test:

   * AST or ALT > Double the normal range limit
   * Total bilirubin > 2.0 mg/dL
   * Ratios of sand dune (eGFR) < 60mL/min/1.73m2
7. Drinking continuously (21 units/week exceeded, 1 unit = 10 g = 12.5 mL of pure alcohol) or who cannot abstain from drinking during clinical trials
8. Those who smoke continuously (more than 10 days) or who cannot quit smoking during the clinical trial period.
9. Those who participated in other clinical or biological equivalence tests within six months prior to the date of the first medication (the last day of the medication for clinical or biological equivalence tests)
10. A person who donated all blood within 60 days prior to the date of the first medication, or who donated the ingredients within 30 days, or who received the blood within 30 days.
11. Those who have taken any prescription or herbal medicine within 14 days prior to the date of the first dose or who have taken any general medication (OTC) within 7 days (however, they may participate in a clinical trial if other conditions are reasonable according to the judgment of the tester.)
12. A person who has taken a medication that induces and inhibits the drug metabolic enzyme, such as barbital drugs, within one month before the start of the test
13. mentally ill and drug addicts
14. A person who has been on a diet (especially grapefruit juice or its products) that can affect the absorption, distribution, metabolism, and excretion of a drug within seven days prior to the date of the first dose.
15. Those who do not agree to exclude the possibility of pregnancy using the medically recognized contraceptives* from the date of the first administration of the clinical trial drug to the date of the last clinical trial medication.

    *Medically accepted contraceptives: intrauterine devices, vascular surgery, intubation and block contraception (male condoms, female condoms, cervical caps, contraceptives, sponges, etc.) or when using a combination of two or more blockage methods.
16. Those who are unwilling or unable to comply with diet and lifestyle guidelines required for clinical testing;
17. Other clinical laboratory tests found that the tester is unfit to participate in a clinical trial due to clinical abnormalities or other reasons (e.g., non-compliance with instructions, non-cooperative attitude, etc.)

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-11-08 (Estimated); Primary Completion 2020-01-08 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic Assessment | 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 and 24hours
  Montelukast and Bepotastine Maximum Plasma Concentration
Pharmacokinetic Assessment | 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 and 24hours
  Montelukast and Bepotastine Area under Curve from time zero to the last quantifiable concentration

SECONDARY OUTCOMES:
Pharmacokinetic Assessment | 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 and 24hours
  Montelukast and Bepotastine Area under Curve from time zero to infinity
Pharmacokinetic Assessment | 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 and 24hours
  Montelukast and Bepotastine time to maximum plasma concentration
Pharmacokinetic Assessment | 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 and 24hours
  Montelukast and Bepotastine half time

CONTACTS AND LOCATIONS:
Overall Officials: Cho Sang Heon, Principal Investigator — Inha University Hospital
Locations (1):
- Inha University Hospital, Junggu, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No